CLINICAL TRIAL: NCT04138706
Title: Initial Vancomycin Taper for the Prevention of Recurrent Clostridium Difficile Infection
Acronym: TAPER-V
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Todd C. Lee MD MPH FIDSA, Associate Professor of Medicine, McGill University; Consultant in Infectious Diseases and Internal Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MP-37-2020-5986
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded placebo-controlled randomized controlled trial:
  A double blind and placebo will be used because the knowledge of being on active drug might influence patient reporting on gastrointestinal symptoms or physician interpretation of such symptoms leading to asymmetrical workup of CDI recurrence and hence bias in the results.
  To avoid other sources of bias post-randomization, patients, research personnel, investigators, endpoint adjudicators, and study analysis will all remain blinded to the intervention status until completion of the analysis and reporting of results. Analysis will be performed by intention to treat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Placebo (Placebo Comparator): Following a 14-day initial vancomycin treatment (125mg QID x14 days), the participant will receive a placebo for an additional 14 days (twice a day x 7 days, then once a day for 7 days).
  Interventions: Drug: Placebos
- Intervention: Extended vancomycin regimen (Active Comparator): Following a 14-day initial vancomycin treatment (125mg QID x14 days), the participant will receive active vancomycin for an additional 14 days (125mg twice a day x 7 days, then 125mg once a day for 7 days).
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Extension of initial vancomycin regimen for the treatment of C. diff from 14 days to 28 days (i.e. an additional 14 days of vancomycin treatment)
  Arms: Intervention: Extended vancomycin regimen
Drug: Placebos — Initial vancomycin treatment (x14 days) will be followed by 14 days of placebo.
  Arms: Control: Placebo

SUMMARY:
The first line therapy for an initial episode of CDI (Clostridium difficile infection) is 10-14 days of oral vancomycin which is now recommended over metronidazole in the 2018 guidelines from the Association of Medical Microbiologists and Infectious Diseases of Canada (AMMI). Although response rates for the treatment of a first episode of CDI now approach 90%, approximately 25% of patients who have a complete response will develop recurrence (rCDI) within 8 weeks. Doctors' ability to predict recurrence is evolving, but remains very limited.

The investigators hypothesize that by extending initial vancomycin therapy with a 2-week tapering regimen this will reduce the risk of rCDI. Starting at the end of the initial 14 days of therapy, participants will be randomized to receive an additional 14-days of placebo or vancomycin taper (125 mg orally twice daily x 7 days followed by 125 mg orally once daily x 7 days). This taper was chosen as it represents two steps of a commonly used 4-week vancomycin taper.

The investigators' proposal to evaluate the extension of initial treatment from 14 to 28 days with a tapering dose of vancomycin represents a practical clinical trial that capitalizes on oral vancomycin's safety profile, worldwide availability, and relatively low cost.

DETAILED DESCRIPTION:
STUDY POPULATION

This is a multi-centre study involving institutions in British Columbia, Ontario, Quebec and Newfoundland. The study population will be drawn from patients cared for as inpatients or outpatients at the participating hospitals. Such patients will have a test positive for C. difficile and will be receiving treatment. The trial will involve only adult patients 18 years of age and older.

Criteria for Recruitment

The microbiology laboratory will notify the study team about a positive CDI test via telephone, email, or fax. The nature of recruitment will then depend on the inpatient status of the patient at the time of the test.

Inpatients:

Pre-existing approval for approaching patients for this study will be obtained from the relevant department heads. The study team will speak with a member of the inpatient treating team (resident physician or faculty physician as appropriate) to determine if the patient is appropriate for recruitment. If this seems to be the case, the patient's file will be rapidly screened to determine eligibility and if the patient is eligible they will be approached for consent.

Outpatients:

The physician who ordered the C. difficile test will be contracted to determine if the patient is appropriate for recruitment. At the invitation of this physician, the investigators will then contact the patient via telephone to evaluate suitability for inclusion and arrange an intake visit.

RANDOMIZATION

For patients who have enrolled in the study, randomization will occur centrally at McGill via an existing internet application and will be performed by permuted block with randomized block sizes. This randomization will be stratified for first episode or first recurrence at study entry to ensure these factors are properly balanced.

TRIAL SCHEDULE

* Day 1: Patient diagnosed with C. difficile and started on standard of care oral vancomycin treatment -> Determine eligibility and obtain permission for approach
* Day 7-10 (Patient's C. difficile has improved and meets eligibility): Consent obtained; randomization; distribution of study drug for day 15 start -> Collection of demographics
* Day 15-28 -> Receipt of study therapy
* Day 28: In person or remote visit
* Day 56: In person or remote visit -> Primary outcome determined, quality of life questionnaire
* Day 90: Study ends for the patient -> Secondary outcomes can be determined
* weekly until Day 56: Brief questionnaire -> By email/text/phone
* biweekly after Day 56: Brief questionnaire -> By email/text/phone
* Ad hoc: If patient has symptoms of recurrence of C. difficile -> Review by ID physician in clinic if possible, otherwise usual doctors or emergency room

Patients will be able to come be assessed for potential relapse by infectious diseases physicians at each site (who may or may not be a part of the study) or could see their usual doctors.

SAMPLE SIZE AND STATISTICAL METHODS

The initial estimates were a risk of recurrence in the control group of 25% and in the intervention group of 15%. With 80% power and an overall alpha of 0.05, it would require 496 patients (rounded to 500) to demonstrate superiority.

After the recruitment of 50 patients, the analytic plan was modified to use a Bayesian framework on April 3rd, 2023, prior to completion of study enrolment and before data were locked and blinded for analysis. This was done to allow for earlier stopping while preserving the overall type 1 error rate and maximal sample size in response to an update to the Infectious Diseases Society of America guidelines for the treatment of C. difficile, which were changed to recommend fidaxomicin as first line therapy in place of vancomycin.

We used adaptR to simulate 50,000 2-armed trials under both the null and alternative hypotheses using the funded 500 patient sample size and interim analyses at 125, 250 and 500 patients. The thresholds for superiority (relative risk <1) were 99% at the first analysis and 97.5% at subsequent analyses. A futility analysis was included whereby the trial would be stopped if there was less than a 15% probability of at least a 4% absolute risk reduction (number needed to treat, NNT ≤ 25). These simulations estimated an overall type 1 error rate of 5.1% with 72.6% power and a median expected sample size of 250 patients.

All binary outcomes were analysed using a Bayesian Generalised Linear Model (binomial family, log link) which yields log relative risk (RR) with 95% Bayesian credible intervals (CrI). These were exponentiated to give risk ratios. Priors were minimally-informative [N~ (0,100)]. Stratification was included in the model and we ran 4 chains of 50,000 Markov Chain Monte Carlo simulations.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients (inpatients and outpatients) who have a treated first episode or first recurrence of CDI.
* CDI will be defined by a positive PCR for toxin gene and/or detection of toxin by EIA or CCA along with three or more episodes of diarrhea within 24 hours
* Patients with a positive test with less than three bowel movements may be included if they initially presented with ileus or if they had pseudomembranous colitis visualized on colonoscopy

Exclusion Criteria:

* Clinical:

  1. Toxic megacolon at presentation not resolved by day 10
  2. For the current episode of CDI: use of metronidazole monotherapy*, fidaxomicin, fecal microbiota transplant or intravenous immunoglobulins

     *Participants may be eligible if they are initially treated with metronidazole but switch to oral vancomycin within 3 days (i.e. maximum 3 days of metronidazole monotherapy).
  3. Previous or current colectomy
  4. Severe allergy/intolerance to oral vancomycin
  5. Patient is expected to die within 3 months from another disease or is expected to be admitted to a palliative care unit
  6. Failure to achieve clinical cure (as above) by day 10
  7. More than 2 episodes of C. difficile in the last 5 years.
  8. Documented history of sensorineural hearing loss (other than presbycusis and noise induced hearing loss). The following patients with documented previous subtypes of sensorineural hearing loss will be excluded from the trial: Menière's disease, multiple sclerosis affecting auditory nerves, otic syphilis, viral cochleitis, autoimmune disorders, previous drug induced hearing loss, and otherwise unexplained sudden sensorineural hearing loss (SSNHL)
  9. Known pregnancy or planning to become pregnant during the study period
  10. Women who are breast feeding
* Administrative:

  1. Expected transfer to a palliative care unit or non-study hospital;
  2. No provincial health insurance
  3. Previously enrolled
  4. No reliable means of outpatient contact
  5. Incompetent without healthcare proxy
  6. Patient stated inability to come to follow up appointments.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
CDI recurrence | Within 56 days of initial vancomycin treatment start date
  Patients will be contacted via text message, email, or phone call weekly until day 56 to determine if they have had a recurrence. After day 56 this will be bi-weekly until day 90.
  Recurrence will be assessed by clinical record review (chart, laboratory, pharmacy records) and direct patient interview. Blinded case summaries will be reviewed in duplicate with disagreement resolved by consensus.
  CDI recurrence will be defined by three or more diarrheal stools/24-hour period coupled with a positive PCR for toxin gene or and/or detection of toxin by EIA or CCA and administration of treatment. However, to avoid missing severe recurrences: for cases of ileus, toxic megacolon, or pseudomembranous colitis on colonoscopy the test result will be used in the absence of three or more stools.

SECONDARY OUTCOMES:
Early recurrence of CDI | Up to day 38 following initial vancomycin start date
  As per primary outcome, at the same duration of follow up as the fidaxomicin registrational trials to allow direct comparison.
Late CDI recurrence | Up to 90 days following initial vancomycin treatment start date
  same as primary outcome
Use of fidaxomicin | Within 90 days of initial vancomycin treatment start date
Number of patients with colectomy | Within 90 days of initial vancomycin treatment start date
Number of patients with fecal microbiota transplantation | Within 90 days of initial vancomycin treatment start date
Number of patient deaths (All-cause death) | Within 90 days of initial vancomycin treatment start date
  If a patient misses their day 28 or day 56 in-person follow up, we will initially review their hospital file to see if they have died. If this does not show death, we will contact the patient (or their proxy) by telephone to determine why they missed the follow up and reschedule it as required. If we cannot reach the patient or their proxy, and the patient has not been replying to the email/text/phone surveys we will search the obituaries.
  After day 56 we will use the survey responses as proof of life. If there is no response to the day 90 survey by day 95, we will first check the hospital file to see if they have died. Then, if vital status is not clear, we will search the obituaries. Then if vital status is still not clear, we will attempt to reach the patient by telephone. If we cannot reach the patient, we will record that patient as lost to follow up but include a sensitivity analysis including these patients as having died.
Emergency Department Visit or Readmission to Hospital | Within 90 days of initial vancomycin treatment start date
  Within 90 days post enrolment we will access the medical record and we will also analyze patient emails/text surveys for all hospital readmissions and will record the date of the first hospital readmission. Patient charts will also be flagged for immediate review should they be readmitted to study centres to assess for the primary and other secondary outcomes. With explicit written patient consent, medical records from outside hospitals will also be requested for review if they report presenting elsewhere.
C. diff associated quality of life | At day 56 after initial vancomycin treatment start date
  At day 56 patients will be asked to provide a measure of self-reported quality of life using the Cdiff32 score which was developed and validated to evaluate health-related quality of life in patients with C.difficile.
  Each item in the Cdiff32 Quality of Life Questionnaire is scored between 0 (worst quality of life) to 100 (best quality of life).
Discontinuation of study drug | At day 28 after initial vancomycin treatment start date
  At the day 28 visit we will inquire about adherence and the quantity of pills remaining.
Receipt of non-study antibiotics | Within 90 days of initial vancomycin treatment start date
  Exposure to antibiotics for infections other than C. difficile may occur. We will ask patients to contact us if this occurs so that the appropriate data can be recorded to account for these effects outside of the study.
Use of off-study vancomycin secondary prophylaxis up to day 90 | Within 90 days of initial vancomycin treatment start date
  Exposure to antibiotics for other infections may lead to the receipt of vancomycin secondary prophylaxis in that context. We will ask patients to contact us if this occurs so that the appropriate data can be recorded to account for these effects outside of the study. If vancomycin secondary prophylaxis has occurred prior to day 28, the patient will stop the study drug to avoid excess vancomycin exposure and this will be recorded.
Safety and tolerability of the vancomycin extension/taper treatment period | Days 15-28 of vancomycin treatment
  We will create a survey at day 28 asking participants to communicate any side effects from the study medication, with a section for detailing any adverse reactions.
Economic analysis | Cost of health care utilization up to 90 days after initial vancomycin treatment start date
  Economic analysis will be carried out from the perspective of the McGill University Health Centre (MUHC) following established guidelines and will be generalized to the rest of Canada.
  We will estimate the average cost per patient of using the interventions under study routinely in patients with C. difficile diarrhea. We will also gather information on the cost of health services use (hospitalizations and other interventions such as colectomy) following this intervention to determine the budget impact compared with routine practice. If the intervention proves efficacious, we will carry out a cost-benefit or cost-effectiveness analysis to determine the incremental cost per case of C. difficile diarrhea avoided. The base case will be the placebo group, to which the treatment will be compared. Further, we will carry out a cost utility analysis to report the incremental cost per unit increase in quality of life as measured by the Cdiff32 score.

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD, MPH, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Emily G McDonald, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (12):
- Canada (12):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre - Eastern Health, St. John's, Newfoundland and Labrador
  - Kingston Health Sciences Centre, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - St Joseph's Health Care, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre (Royal Victoria Hospital), Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
We will conform to our institutional policies and the policy of the accepting journal.

REFERENCES:
- [Background] Leffler DA, Lamont JT. Clostridium difficile infection. N Engl J Med. 2015 Apr 16;372(16):1539-48. doi: 10.1056/NEJMra1403772. No abstract available. PMID 25875259
- [Background] Lessa FC, Gould CV, McDonald LC. Current status of Clostridium difficile infection epidemiology. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S65-70. doi: 10.1093/cid/cis319. PMID 22752867
- [Background] Levy AR, Szabo SM, Lozano-Ortega G, Lloyd-Smith E, Leung V, Lawrence R, Romney MG. Incidence and Costs of Clostridium difficile Infections in Canada. Open Forum Infect Dis. 2015 Jun 3;2(3):ofv076. doi: 10.1093/ofid/ofv076. eCollection 2015 Sep. PMID 26191534
- [Background] Dobson G, Hickey C, Trinder J. Clostridium difficile colitis causing toxic megacolon, severe sepsis and multiple organ dysfunction syndrome. Intensive Care Med. 2003 Jun;29(6):1030. doi: 10.1007/s00134-003-1754-7. Epub 2003 May 7. No abstract available. PMID 12734650
- [Background] Mylonakis E, Ryan ET, Calderwood SB. Clostridium difficile--Associated diarrhea: A review. Arch Intern Med. 2001 Feb 26;161(4):525-33. doi: 10.1001/archinte.161.4.525. PMID 11252111
- [Background] McDonald EG, Milligan J, Frenette C, Lee TC. Continuous Proton Pump Inhibitor Therapy and the Associated Risk of Recurrent Clostridium difficile Infection. JAMA Intern Med. 2015 May;175(5):784-91. doi: 10.1001/jamainternmed.2015.42. PMID 25730198
- [Background] Sheitoyan-Pesant C, Abou Chakra CN, Pepin J, Marcil-Heguy A, Nault V, Valiquette L. Clinical and Healthcare Burden of Multiple Recurrences of Clostridium difficile Infection. Clin Infect Dis. 2016 Mar 1;62(5):574-580. doi: 10.1093/cid/civ958. Epub 2015 Nov 17. PMID 26582748
- [Background] Rodrigues R, Barber GE, Ananthakrishnan AN. A Comprehensive Study of Costs Associated With Recurrent Clostridium difficile Infection. Infect Control Hosp Epidemiol. 2017 Feb;38(2):196-202. doi: 10.1017/ice.2016.246. Epub 2016 Nov 7. PMID 27817758
- [Background] Olsen MA, Yan Y, Reske KA, Zilberberg MD, Dubberke ER. Recurrent Clostridium difficile infection is associated with increased mortality. Clin Microbiol Infect. 2015 Feb;21(2):164-70. doi: 10.1016/j.cmi.2014.08.017. Epub 2014 Oct 12. PMID 25658560
- [Background] The Lancet. A new approach to treating infection. Lancet. 2018 Feb 24;391(10122):714. doi: 10.1016/S0140-6736(18)30320-9. No abstract available. PMID 29486930